CLINICAL TRIAL: NCT00824395
Title: Mitochondria and Metabolic Syndrome in a Southern California Chinese Cohort
Brief Title: The Genetics of Diabetes in Southern California Chinese Americans
Status: Withdrawn | Type: Observational
Why Stopped: Non applicable clinical trial
Sponsor: University of California, Irvine (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-4675
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes; Metabolic Syndrome
Keywords: diabetes; type 1; type 2; metabolic syndrome; mitochondria
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Individuals with diabetes
- 2: Individuals without diabetes

SUMMARY:
The purpose of this research study is to investigate the genetic causes of diabetes. Specifically, we are interested in the mitochondrial genome and how variants in the mitochondrial genome influence a person's risk to develop diabetes and metabolic syndrome.

DETAILED DESCRIPTION:
Since our laboratory's initial linkage of Type 2 diabetes to a mtDNA rearrangement in a three generation maternal pedigree 13 years ago, there has been increasing support for our hypothesis that mitochondrial dysfunction plays an important role in the etiology of Type 2 Diabetes Mellitus (DM) and the overlapping Metabolic Syndrome (MS). With this study we are planning an extensive investigation of defects in mitochondrial oxidative phosphorylation (OXPHOS) caused potentially by deleterious sequence variants in the mitochondrial DNA (mtDNA). As the primary objective we are trying to further substantiate 2 hypotheses: 1) that these diabetogenic mtDNA variants, which are proposed to range from recent, relatively severe, mutations will result in substantial OXPHOS defects with familial DM & MS and 2) that ancient, relatively mild polymorphisms result in partial OXPHOS defects and an increase in the risk to develop DM & MS.

ELIGIBILITY:
Inclusion Criteria:

* Chinese or Taiwanese ancestry
* Resident of Southern California
* Age between 40 and 65
* Both people with and without diabetes are welcome to enroll.

Exclusion Criteria:

* Younger than 40 years or older than 65 years
* Ancestry is not Chinese or Taiwanese
* Not a resident of Southern California

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are currently recruiting Chinese Americans living in Southern California, espcially in Orange and Los Angeles Counties. We are particularly in need of Chinese American men and women with diabetes as well as healthy male controls. We can arrange for offsite weekend trips to cities within LA or Orange Counties for eligible groups of 10 or more people.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Wallace, PhD, Principal Investigator — UC Irvine Center for Mitochondrial Medicine
Locations (1):
- UC Irvine General Clinical Research Center, Irvine, California, United States